CLINICAL TRIAL: NCT05019027
Title: N-of-1 Trials to Promote Deprescribing in Older Adults With Transthyretin Cardiac Amyloidosis
Brief Title: N-of-1 for Beta-Blockers in Cardiac Amyloidosis
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: U.S. Deprescribing Research Network (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-07023710
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Cardiac Amyloidosis; Heart Diseases; TTR Cardiac Amyloidosis
Keywords: beta blocker; cardiac amyloidosis; HFpEF; deprescribing; heart failure
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Heart Diseases; Heart Failure | interventions — Adrenergic beta-Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- On-Off Sequence (Other): This arm will follow an On-Off sequence. This is the only arm in the study. Subjects will begin in the On phase (Period 1), where they will be on their beta-blocker (or the highest dose they can safely tolerate) as previously prescribed to the subjects by their physician. Subjects will then continue to the Off phase (Period 2) where they will down-titrate their beta-blocker by 50% each week until they are completely off the drug (or the lowest dose they can safely tolerate) for a total of two weeks. At the end of Period 2, the subjects will have their End of Intervention visit to determine if they would like to continue or discontinue their beta-blockers for the foreseeable future.
  Interventions: Drug: Beta blocker

INTERVENTIONS:
Drug: Beta blocker — The intervention is a single-arm crossover withdrawal/reversal design (On vs Off) with 2 total periods, each period lasting between up to 6 weeks. During the On period, subjects will be on their beta blocker. During the Off period, their beta blockers will be down-titrated by 50% each week and until subsequently discontinued (or the lowest dose the subject can safely tolerate).
  Other Names:
  * acebutolol
  * atenolol
  * betaxolol
  * bisoprolol
  * carvedilol
  * labetalol
  * metoprolol succinate
  * metoprolol tartrate
  * nadolol
  * nebivolol
  * penbutolol
  * pindolol
  * propranolol

SUMMARY:
The study team will generate preliminary data on whether patients with cardiac amyloidosis feel better when their beta-blocker is stopped. To achieve this objective, 20 N-of-1 trials (on vs. off) will be conducted, and the study team will subsequently interview participants to better understand their outcomes. Each subject will participate in 2 periods lasting between up to 6 weeks each based on each patient's health profile. We will also engage stakeholders to understand the acceptability and feasibility of deprescribing N-of-1 trials. The N-of-1 trials will be iteratively refined in real-time based on feedback.

DETAILED DESCRIPTION:
The intervention is an unblinded NIH Stage I of Behavioral Intervention Development trial, using a single-arm crossover withdrawal/reversal design (On [A] vs. Off [B]) with 2 periods, each period lasting up to 6 weeks, allowing for down-titration and washout. During the On (A) period, participants will be on their beta-blocker (or the highest dose they can safely tolerate), as previously prescribed to the subjects by their physician. During the Off (B) period, their beta-blockers will be down-titrated and subsequently discontinued (or at the lowest dose they can safely tolerate); we will decrease the dose of beta-blocker by 50% every week regardless of which beta-blocker they are on, similar to an algorithm used in a prior deprescribing trial.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory adults age ≥65 years with TTR-cardiac amyloidosis (confirmed by PYP scan or biopsy)
2. Taking beta-blocker

Exclusion Criteria:

1. Other compelling indication(s) for beta-blockers:

   1. Angina
   2. Acute coronary syndrome, myocardial infarction or coronary artery bypass surgery in prior 3 years
   3. Atrial arrhythmia with hospitalization for rapid ventricular response, prior 1 year
   4. Heart rate >100 bpm within the prior 3 months
   5. Atrial arrhythmia with ventricular rate >90 beats per minute within the prior 3 months
   6. Systolic blood pressure readings >160 mmHg within the prior 1 month, unless classified as white coat hypertension/effect (e.g., migraine prevention, anxiety symptom management, hyperthyroidism, essential tumor reduction)
2. Clinical instability (N-of-1 trials are appropriate for stable conditions only)

   1. Decompensated heart failure
   2. Hospitalized in the past 30 days
   3. Medication changes or procedures in the prior 14 days that could confound observations/data at Principal Investigator discretion
   4. Anticipated medication changes or procedures in subsequent 3 months that could confound observations/data at PI discretion
   5. Clinical instability from other medical issues
3. Estimated life expectancy <6 months
4. Moderate-severe dementia or psychiatric disorder precluding informed consent
5. Language barrier that will preclude informed consent and ability to comprehend study procedures
6. Non-compliance or inability to complete study procedures
7. Enrollment in a clinical trial not approved for co-enrollment
8. Any condition that, in Principal Investigator or treating physician's opinion, makes the patient unsuitable for study participation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The change in exercise capacity when on beta-blocker versus when off beta-blocker, as measured by peak oxygen consumption (VO2) during Cardiopulmonary Exercise Test (CPET). | End of Period 1 (Week 2, 3, 4, 5, or 6) and Period 2 (Week 8, 9, 10, 11, or 12)
  To understand the changes in exercise capacity between the On and Off phase via a Peak oxygen consumption (VO2) Cardiopulmonary Exercise Test. Cardiopulmonary exercise testing (CPET) measures breath-by-breath oxygen production during symptom-limited exercise on a stationary bike or treadmill. This permits calculation of peak oxygen consumption (VO2). Percent predicted peak VO2 for body weight will also be calculated.
The change in patient-reported health status when on beta-blocker versus when off beta-blocker, as measured by Kansas City Cardiomyopathy Questionnaire (KCCQ-12). | Baseline, End of Period 1 (Week 2, 3, 4, 5, or 6), End of Period 2 (Week 8, 9, 10, 11, or 12)
  The Kansas City Cardiomyopathy Questionnaire (KCCQ-12) is a heart failure-specific health status survey. Questions are ranked on 5- to 7-point Likert scales, with higher scores indicating better health status.
The change in patient-reported quality of life when on beta-blocker versus when off beta-blocker, as measured by the EuroQol-5d Visual Analogue Scale. | Baseline; End Period 1 (Weeks 2, 3, 4, 5, or 6), End of Period 2 (Weeks 8, 9, 10, 11, or 12)
  The EuroQol-5D Visual Analogue System (EQ-5D VAS) indicates patient-perceived health on a vertical visual analogue scale. The scale ranges from 0, indicating poorest health, to 100, indicating best health.

SECONDARY OUTCOMES:
Change in patient-reported quality of life when on beta-blocker, as measured by the Patient-Reported Outcome Measurement Information System-29 (PROMIS-29) | Baseline; Weekly for up to 12 weeks; End of Period 1 (Week 2, 3, 4, 5, or 6), Period 2 (Week 8, 9, 10, 11, or 12)
  Patient-Reported Outcome Measurement Information System-29 (PROMIS-29) is a health-related quality of life survey, with questions from 6 domains: depression, anxiety, physical function, pain interference, sleep disturbance, and ability to engage in social roles and activities. Questions are ranked on a 5-point Likert scale, with higher scores at times indicating better quality of life, and at other times indicating poorer quality of life. There is a pain rating scale ranging from 0 to 10, with higher scores indicating higher pain level. Scores are reported for each domain, as well as for pain rating.

CONTACTS AND LOCATIONS:
Overall Officials: Parag Goyal, MD, MSc, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No